CLINICAL TRIAL: NCT04700254
Title: The Effect of COVID-19 National Lockdown on People With Diabetes Mellitus Regarding Their Anxiety, Depression and Eating Attitudes, in Relation to Adjusted Work and Family Conditions
Brief Title: Anxiety, Depression and Eating Attitudes of Diabetes Mellitus Patients During COVID-19 Lockdown in Greece
Status: Completed | Type: Observational
Sponsor: Chania General Hospital "St. George" (Other)
Collaborators: AHEPA University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Diabetes and COVID-19
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus; SARS-CoV-2
Keywords: Diabetes Mellitus; Anxiety; Depression; Eating attitudes
MeSH Terms: conditions — Diabetes Mellitus; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- working condition: In order to further explore the differences among working status the data will be categorized into three different groups: suspension of work, employment and unemployment.
  Interventions: Other: DASS questionnaire; Other: EAT-26 questionnaire
- Family status: In order to xplore the differences among the family status, the data will be categorized into the married and the singles DM patients.
  Interventions: Other: DASS questionnaire; Other: EAT-26 questionnaire
- BMI status: In order to further explore BMI scale results, we divided the data obtained from the participants into normal (18.50 - 24.99 kg/m2), overweight (25-29.99 kg/m2) and obese (≥30 kg/m2), according to the international classification of the World Health Organisation (WHO).
  Interventions: Other: DASS questionnaire; Other: EAT-26 questionnaire

INTERVENTIONS:
Other: DASS questionnaire — The DASS is a 42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress
Other: EAT-26 questionnaire — The Eating Attitudes Test (EAT-26), is a self-report 26-item questionnaire of symptoms and concerns characteristic of eating disorders.

SUMMARY:
The aim of this observational, cross-sectional study is to evaluate the impact of the second national COVID-19 lockdown in Greece, regarding the aspects of depression, anxiety and eating habits, in relation to the adjusted work and family conditions, among diabetes mellitus patients.

DETAILED DESCRIPTION:
The national Lockdown was an attempt by the Governments around the world to prevent the spreading of the SARS-CoV-2. This pandemic turned out to be a major public health challenge. In Greece two national lockdown were imposed in 2020, among other measures, in order to minimize the spread of the SARS-CoV-2. The national lockdown consists of the temporary closure of the sports arenas, theaters, cafeterias, restaurants, cinemas, archaeological sites, schools, churches universities and most of the businesses . The first national lockdown in Greece was imposed from March 23th to May 4th and the second one took place from November 6th until now. Such a lockdown that forces the majority of individuals to stay at home for a prolonged period of time, except the controlled movement of the individuals for some cases, could expectedly enough have quite an impact on the daily life of people with diabetes mellitus. Changes to dietary habits, limitation of physical activity, as well as the psychological aspects like those of depression and anxiety have been detected. The aim of this study is to evaluate the impact of the second national lockdown in Greece, regarding the aspects of depression, anxiety and eating habits, in relation to the adjusted work and family conditions, among diabetes mellitus patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* Type 1 Diabetes Mellitus
* Type 2 Diabetes Mellitus
* MODY Diabetes Mellitus

Exclusion Criteria:

* age <18 years
* gestational Diabetes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from the outpatient diabetes clinic of General Hospital of Chania and the Diabetes Center of the1st Propaedeutic Department of Internal Medicine of AHEPA General University Hospital of Thessaloniki in Greece. All participants prior to completing the survey had to give their informed consent in order to continue. Participants were free to abandon the survey at any time without any sanctions.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
DASS (Depression) | Time Frame: Brief standardised questionnaire not exceeding 8 minutes. Administered during the data collection phase, no intervention involved, this is a cross-sectional observation study.
  Minimum score 0 maximum score 42 of the depression subscale of the DASS questionnaire Higher scores mean a worse outcome
DASS (Anxiety) | Time Frame: Brief standardised questionnaire not exceeding 8 minutes. Administered during the data collection phase, no intervention involved, this is a cross-sectional observation study.
  Minimum score 0 maximum score 42 of the anxiety subscale of the DASS questionnaire Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Eating Attitudes Test (EAT-26) | Time Frame: Brief standardised questionnaire not exceeding 8 minutes. Administered during the data collection phase, no intervention involved, this is a cross-sectional observation study.
  Minimun score 0 maximum score 78 Scores greater than 20 indicate a need for further investigation by a qualified professional.
  Low scores (below 20) can still be consistent with serious eating problems.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Chania, Chania, Crete, Greece

IPD SHARING:
Plan to Share IPD: Undecided
contact via e-mail

REFERENCES:
- [Result] Aragona M, Rodia C, Bertolotto A, Campi F, Coppelli A, Giannarelli R, Bianchi C, Dardano A, Del Prato S. Type 1 diabetes and COVID-19: The "lockdown effect". Diabetes Res Clin Pract. 2020 Dec;170:108468. doi: 10.1016/j.diabres.2020.108468. Epub 2020 Sep 25. PMID 32987040
- [Result] Sakelliadis EI, Katsos KD, Zouzia EI, Spiliopoulou CA, Tsiodras S. Impact of Covid-19 lockdown on characteristics of autopsy cases in Greece. Comparison between 2019 and 2020. Forensic Sci Int. 2020 Aug;313:110365. doi: 10.1016/j.forsciint.2020.110365. Epub 2020 Jun 12. PMID 32563134
- [Result] Sidor A, Rzymski P. Dietary Choices and Habits during COVID-19 Lockdown: Experience from Poland. Nutrients. 2020 Jun 3;12(6):1657. doi: 10.3390/nu12061657. PMID 32503173
- [Result] Ruiz-Roso MB, Knott-Torcal C, Matilla-Escalante DC, Garcimartin A, Sampedro-Nunez MA, Davalos A, Marazuela M. COVID-19 Lockdown and Changes of the Dietary Pattern and Physical Activity Habits in a Cohort of Patients with Type 2 Diabetes Mellitus. Nutrients. 2020 Aug 4;12(8):2327. doi: 10.3390/nu12082327. PMID 32759636
- [Result] Pellegrini M, Ponzo V, Rosato R, Scumaci E, Goitre I, Benso A, Belcastro S, Crespi C, De Michieli F, Ghigo E, Broglio F, Bo S. Changes in Weight and Nutritional Habits in Adults with Obesity during the "Lockdown" Period Caused by the COVID-19 Virus Emergency. Nutrients. 2020 Jul 7;12(7):2016. doi: 10.3390/nu12072016. PMID 32645970